CLINICAL TRIAL: NCT06041841
Title: A Phase 2, Single-arm, Open-label Study to Assess Efficacy and Safety of LB54640 in Patients With Obesity Due to POMC, PCSK1, or LEPR Deficiency.
Brief Title: A Phase 2 Study to Assess Efficacy and Safety of LB54640 in Patients With Genetic Obesity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-MCCL004
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: POMC Deficiency Obesity; PCSK1 Deficiency Obesity; LEPR Deficiency Obesity

STUDY DESIGN:
Intervention Model Description: This is a study where each participant participates for up to 56 weeks. The study consists up to 7 visits to study center which include a Screening period, treatment period, and a follow-up period. Eligible participants who are willing to enter the long-term extension period and who are judged by the study doctor to have no safety concerns, will continue to receive LB54640 at the same dose level from the treatment period. The long-term extension period will be followed by a follow-up period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- POMC/PCSK1/LEPR cohort (Experimental): LB54640 once daily by oral administration
  Interventions: Drug: LB54640

INTERVENTIONS:
Drug: LB54640 — LB54640 QD Oral

SUMMARY:
The purpose of the study was to assess the efficacy of LB54640 in participants with rare genetic disorders of obesity

DETAILED DESCRIPTION:
Patients with obesity due to POMC, PCSK1 or LEPR deficiency will be enrolled to receive LB54640 by oral administration for 16 weeks. After 16 weeks of treatment, the participant may enter a long term extension phase and receive treatment for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥12 years at the time of enrollment and diagnosed with genetic obesity due to POMC, PCSK1, or LEPR deficiency mutations.
* Obesity is defined as BMI ≥30 kg/m2 for participants ≥18 years of age or BMI ≥95th percentile for age and gender for participants <18 years of age.

Exclusion Criteria:

* Participants with recent (within 2 months, prior to Screening and up to enrollment) intensive diet/exercise regimen that resulted in >2% weight loss, use of medication to treat obesity (within 3 months of first dose of LB54640 with certain exceptions), or weight loss surgery within 6 months prior to Screening or prior surgery which resulted in >10% weight loss with no evidence of weight regain are excluded
* History of major surgical procedure
* Weight loss surgery within the previous 6 months
* Any history of a suicide attempt, or any suicidal behavior
* HbA1c >10.9%
* Fasting glucose level >270 mg/dL

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of BMI | From baseline to Week 16

SECONDARY OUTCOMES:
Frequency and severity of adverse events (AE) | From first dose up to Week 52
Frequency and severity of adverse events of special interest (AESI) | From first dose up to Week 52
Mean change and mean percentage change from baseline in body weight | From baseline up to Week 52
Mean change and mean percentage change from baseline in waist circumference. | From baseline up to Week 52
Mean change and mean percentage change from baseline in Hunger Questionnaire Scores | From baseline up to Week 52
  The question will asked using the Hunger Questionnaire. The questionnaire consists of a new 5-item, patient-reported scale assessing major eating-related factors (worst and average hunger, appetite, craving, and satiety).
Mean change and mean percentage change from baseline in body composition assessed by dual energy x-ray absorptiometry | From baseline up to Week 52
  Fat mass and lean mass will be measured through dual energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (2):
- Pitié Salpêtrière hospital and Sorbonne Université, Paris, France
- Cambridge university, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No